CLINICAL TRIAL: NCT05106881
Title: Usability and Satisfaction Test to the Wearable Walking-assist Robot (GEMS-H) in the Community-dwelling Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-04-058
Record Dates: First submitted 2021-10-14; First posted 2021-11-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Gait Disorders in Old Age
Keywords: Wearable hip assist robot; Gait; User test; Robot gait training; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training with Gait Enhancing and Motivating System (GEMS-H) Robot (Experimental): Training consists of 15 minutes task-specific training and 20-30 minutes functional gait training on varied environments with device.
  Interventions: Device: Training with Gait Enhancing and Motivating System (GEMS-H) Robot

INTERVENTIONS:
Device: Training with Gait Enhancing and Motivating System (GEMS-H) Robot — Training consists of 15 minutes task-specific training and 30 minutes functional gait training on varied environments with device.
  Other Names: Training with GEMS-H

SUMMARY:
The purpose of this study is to investigate the userbility and satisfaction of one-off functional gait training with the Gait Enhancing and Motivating System-Hip type (GEMS-H) on locomotor function in normal adults including the elderly.

DETAILED DESCRIPTION:
The GEMS-H is a hip-type assist device developed by the Samsung Advanced Institute of Technology. The GEMS-H is worn around the waist and fastened at the waist and thighs by a set of belts with velcro to assist motion at the hip joints. The device weighs 2.1kg, and has 2 brushless direct current motors running on a rechargeable lithium ion battery. The normal operation time for the device is 2 hours. The GEMS-H is available in three sizes to fit various waist/hip sizes: small, medium, and large. The width of each version can be adjusted further to fit individual body size within the circumference range. Also, the thigh frames are available in three sizes (large, medium, and small) for different leg lengths. It is controlled through a custom built application on a hand held tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 40 to less than 85 years without a history of central nervous system disease

Exclusion Criteria:

* Those who have difficulty walking independently due to problems such as visual field defects or fractures
* Those who have difficulty participating in exercise programs due to adult diseases such as uncontrolled hypertension and diabetes
* Those who have difficulty understanding the exercise program due to severe cognitive decline (Korean-Mini-Mental State Examination, K-MMSE≤10)
* Those who are at risk of falling while walking due to severe dizziness
* Those who are less than 140 cm or more than 185 cm in height that is not suitable size for the wearing of the walking assistance robot
* Those who are overweight based on body mass index (BMI) 35 or higher

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test from baseline in gait speed | Baseline, After 45minutes of functional gait training (one-time experience)
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Change in Timed Up and Go test (TUG) from baseline in balance | Baseline, After 45minutes of functional gait training (one-time experience)
  Measure of dynamic balance function. 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Changes in Short Physical Performance Battery (SPPB) from baseline | Baseline, After 45minutes of functional gait training (one-time experience)
  SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Changes in Four Square Step Test (FSST) from baseline | Baseline, After 45minutes of functional gait training (one-time experience)
  FSST is used to assess dynamic stability and the ability of the subject to step over low objects forward, sideways, and backward.
Change in 6 minute walk test (6MWT) from Baseline | Baseline, After 45minutes of functional gait training (one-time experience)
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
User Satisfaction Questionnaire | After 45minutes of functional gait training (one-time experience)
  We evaluate the satisfaction questionnaire for GEMS-H use.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea